CLINICAL TRIAL: NCT04249973
Title: Detection of Metabolite Biomarkers for the Early Diagnosis and Prognosis of Cow's Milk Allergy in Children
Status: Active, not recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201734666
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cow Milk Allergy; Food Allergy
Keywords: Metabolomics; Microbiome analysis
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — Urine and fecal samples will be collected at the family's home. The majority of the patients will only be sampled once. But a small number of patients will be followed-up yearly for 3-4 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IgE-mediated cow's milk allergy: Feces and urine samples are collected by the parents at home. Feces is collected out of the diaper or using a fecotainer. Urine is collected directly or using a urine collection pad. Additionally, the parents fill in a short questionnaire regarding the symptoms of their child, their clinical history and relevant information regarding the development of food allergies.
  Interventions: Other: Collection of urine and feces
- Suspected of cow's milk allergy, but with negative diagnosis: Feces and urine samples are collected by the parents at home. Feces is collected out of the diaper or using a fecotainer. Urine is collected directly or using a urine collection pad. Additionally, the parents fill in a short questionnaire regarding the symptoms of their child, their clinical history and relevant information regarding the development of food allergies.
  Interventions: Other: Collection of urine and feces
- IgE-mediated food allergy, other than cow's milk: Feces and urine samples are collected by the parents at home. Feces is collected out of the diaper or using a fecotainer. Urine is collected directly or using a urine collection pad. Additionally, the parents fill in a short questionnaire regarding the symptoms of their child, their clinical history and relevant information regarding the development of food allergies.
  Interventions: Other: Collection of urine and feces
- Healthy brothers and sisters: Feces and urine samples are collected by the parents at home. Feces is collected out of the diaper or using a fecotainer. Urine is collected directly or using a urine collection pad. Additionally, the parents fill in a short questionnaire regarding the symptoms of their child, their clinical history and relevant information regarding the development of food allergies.
  Interventions: Other: Collection of urine and feces

INTERVENTIONS:
Other: Collection of urine and feces — Urine and feces are collected at the families home. A short questionnaire is filled in by the parents

SUMMARY:
In this study, fecal and urine samples will be collected from children diagnosed with :

* IgE mediated cow's milk allergy,
* suspected of a cow's milk allergy, but with negative diagnosis
* IgE mediated food allergy other than cow's milk
* healthy brothers and sisters of the first three groups A subset of patients with IgE-mediated cow's milk allergy will be asked to provide a urine and fecal sample yearly for prognostic purposes.

The samples will be analyzed using a technique called metabolomics to identify biomarker candidates with diagnostic and/or prognostic potential. Additionally, microbiome analysis will be performed to map the microbiome of all groups.

DETAILED DESCRIPTION:
In this study urine and fecal samples will be collected from children until the age of 4 years old. The metabolome and microbiome of children with IgE mediated cow's milk allergy (1) (CMA) will be compared to that of children in three control groups: (2) children suspected of IgE mediated CMA, but with negative diagnosis, (3) children with an IgE mediated food allergy other than cow's milk and (4) healthy brothers and sisters of the first 3 groups. Children will be divided into these four groups based on the current diagnostic tests, including IgE measurements (skin prick tests and IgE measurements in venous blood samples), clinical history of the patients and their response to elimination diets. Samples will be collected shortly after diagnosis.

In a second phase of this study several patients will be followed up for several years (3 - 4 years), for which yearly a urine and fecal sample will be collected. Children included in this part will be younger than 1 year at the moment of their first sample donation, and diagnosed with IgE mediated CMA. This longitudinal follow-up is based on the microbial difference at the age between 3 to 6 months between children that will have a persistent allergy and the ones that will grow out of their allergy. These differences are anticipated to be translated in to the metabolomes of these children.

The samples will be collected at home and have to be frozen immediately after sample collection, after which they will be picked up by the researchers. The samples will be analyzed using a technique called metabolomics, using UHPLC-HRMS (Ultra-High Performance Liquid Chromatography coupled to High-Resolution Mass Spectrometry). After analysis the metabolic profiles of the different groups will be compared to each other using multivariate statistical analysis. This methodology will be applied to find biomarker candidates with good sensitivity and specificity for future CMA diagnosis or prognosis. Additionally, the identified biomarkers could provide more insights into the mechanisms behind the disease, which can aid in future therapy.

Microbiome analysis will be performed using qPCR and 16S rRNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* IgE mediated cow's milk allergy
* suspected for a cow's milk allergy, but with negative diagnosis (e.g. non-IgE mediated cow's milk allergy)
* IgE mediated food allergy other than cow's milk
* healthy brothers and sisters from the first three groups

Exclusion Criteria:

* children of 5 years or older

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The cohorts will be selected from several hospitals in Flanders (UZ Ghent, AZ Jan Palfijn, AZ Maria Middelares, AZ Sint-Jan, Sint-Vincentius Deinze, UZ Leuven, AZ Nikolaas, ZNA Koningin Paola Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | Samples will be analyzed in the beginning of 2020, the results are expected mid 2020
  Urine and fecal samples will be analyzed using a technique called metabolomics, which analyses all small molecules (metabolites) present in a biological fluid. These metabolites will be used to find biomarkers that are related to the disease and could have diagnostic or prognostic potential. Additionally, these metabolites could give more insights into the development and maintenance of the disease.
Microbiome analysis | Samples will be analyzed mid 2020
  The microbiomes of all groups will be analyzed because it has been described in literature that the microbiome can differ between healthy and allergic individuals. The microbial signatures related with IgE mediated CMA can give more insights into the pathology of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Van Winckel, Prof, Principal Investigator — University Ghent
Locations (8):
- Belgium (8):
  - AZ Sint-Jand, Bruges, Oost-Vlaanderen
  - AZ Sint Vincentius, Deinze, Oost-Vlaanderen
  - AZ Jan Palfijn, Ghent, Oost-Vlaanderen
  - Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Maria Middelares, Ghent, Oost-Vlaanderen
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - ZNA Koningin Paola Kinderziekenhuis, Antwerp

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers